CLINICAL TRIAL: NCT05161754
Title: Tonsillectomy and Risk of Post-tonsillectomy Hemorrhage - a Randomized Clinical Trial
Brief Title: Tonsillectomy and Risk of Post-Tonsillectomy Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Michael F Howitz, Principal Investigator, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-20036864
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Tonsillectomy
MeSH Terms: interventions — Hemostasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment 1 (Experimental): Participants left tonsil: cold dissection and hot hemostasis. Participants right tonsil: cold dissection and cold hemostasis.
  Interventions: Procedure: Hemostasis
- Treatment 2 (Experimental): Participants right tonsil: cold dissection and hot hemostasis. Participants left tonsil: cold dissection and cold hemostasis.
  Interventions: Procedure: Hemostasis

INTERVENTIONS:
Procedure: Hemostasis — Hot hemostasis include bipolar and monopolar diathermy. Cold hemostasis include surgical knotting of the tonsil pillar and compression.

SUMMARY:
Post-tonsillectomy hemorrhage (PTH) is a feared complication to tonsillectomy. Tonsillectomy may be performed using different surgical techniques, which include both "cold" and "hot" dissection and hemostasis - but the technique may have a great impact on the risk of PTH. As of today there is no standard on how to perform hemostasis during tonsillectomy in Denmark.

The aim of this study is to clarify whether cold dissection with either cold or hot hemostasis during the surgical procedure of tonsillectomy holds the lowest risk of PTH. Secondary objective is to address whether there is a difference in pain perception associated with the two procedures. The null hypothesis is that there is no difference in PTH between cold and hot hemostasis in tonsillectomy.

DETAILED DESCRIPTION:
Tonsillectomy is one of the most common procedures in the field of otorhinolaryngology, and in 2012 the yearly incidence was 129,4 per 100.000 inhabitants in Denmark. One feared complication among patients as well as physicians is post-tonsillectomy hemorrhage (PTH). The PTH incidence varies between 0,5 to 33 procent in reported studies, and an increased incidence from 1991 to 2012 has been showed in a Danish study.

PTH is in the literature typically divided into a primary PTH occurring within 24 hours of tonsillectomy and a secondary PTH occurring in a bell-shaped incidence curve from day one after tonsillectomy to normally no risk 14 days after tonsillectomy when the tonsil eschar is discharged, and the tonsil bed is healed. The highest incidence of PTH is on day 0 and day 6.

The risk of PTH has been studied for the different surgical techniques. Both dissection and hemostasis may be performed by a "cold" or "hot" procedure, with the latter referring to the use of a heated instrument (coblation, diathermy, harmonic scalpel, various lasers ect.).

Cold dissection with no heated hemostasis is associated with the overall lowest risk of delayed PTH in a Swedish study. They showed that the risk of delayed PTH increases with the use of a bipolar diathermy for dissection and further increased if used for hemostasis in the tonsil bed.

A multicenter study from England and Northern Ireland found an over-all risk of PTH at 3.3 procent. The highest risk of PTH was found when hot technique was applied for both dissection and hemostasis, the relative risk of PTH was 3.1, comparing to a relative risk of 2.2 when dissection was conducted with cold steel and diathermy. Reference was cold steel tonsillectomy alone. Coblation held the highest risk (3.4).

A review article from 2019 on ten published articles (n=3,987) concludes that suturing tonsil pillars after tonsillectomy may be beneficial to lower PTH after cold tonsillectomy. Five studies looked at postoperative pain reduction after tonsil pillar suturing and the conclusion is that this will likely need further investigation, as there are many factors that can influence pain perception. The operation time increased with in average eight minutes when performing suture on the tonsil pillar, basis and/or bed.

In Denmark there is no standard on how to perform hemostasis during tonsillectomy. It is up to the surgeon to choose. In Denmark anno 2020 and at least the past two decades the preferred techniques have been cold dissection of the tonsil, some use knotting of the tonsil pillar, while other use diathermy on the tonsil pillar and most perform secondary hot diathermy of the tonsil bed to acquire hemostasis per-operatively.

Randomized clinical trials are regarded as the best way to study the safety and efficacy of a treatment. To our knowledge, from search at Pubmed.gov, clinicaltrials.gov and clinicaltrialsregister.eu a similar study has not been conducted and no similar study is registered undergoing elsewhere. Following, we would like to initiate this randomized clinical trial to clarify which hemostasis procedure has the overall lowest risk of PTH. Results from a study like this will be important scientific input in an ongoing discussion among Ear, nose and throat doctors and of beneficial for future patients undergoing tonsillectomy.

In short, the surgeon is randomly instructed to conduct normal procedure (cold dissection and bipolar diathermy) on one tonsil, and on the other tonsil use cold dissection and cold hemostasis (surgical knotting of the tonsil pillar and compression). Our endpoints are primary and secondary PTH and pain perception.

ELIGIBILITY:
Inclusion Criteria:

All patients at the age of 12 years or older referred for tonsillectomy from a medical doctor will be asked to participate.

Exclusion Criteria:

* Patients under the age of 12 years.
* If using prescriptive anticoagulations.
* If known with a coagulopathy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Number of bleeding episodes | Postoperative day 0 to 30
  Number of bleeding episodes from each tonsilbed.

SECONDARY OUTCOMES:
Pain perception | Postoperative day 0 to 30
  Pain Scores on the Visual Analog Scale (VAS)- for the left and right throat side respectively. The VAS ranges from 0 to 10, with 0 indicating no pain and higher scores indicating greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frantz Howitz, MD, PhD, Principal Investigator — North Zealand University Hospital
Locations (2):
- Denmark (2):
  - Charlottenlund Privat Hospital, Charlottenlund
  - Nordsjaellands Hospital, Hillerød

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juul ML, Rasmussen ER, Rasmussen SHR, Sorensen CH, Howitz MF. A nationwide registry-based cohort study of incidence of tonsillectomy in Denmark, 1991-2012. Clin Otolaryngol. 2018 Feb;43(1):274-284. doi: 10.1111/coa.12959. Epub 2017 Sep 13. PMID 28851039
- [Background] Kvaerner KJ. Benchmarking surgery: secondary post-tonsillectomy hemorrhage 1999-2005. Acta Otolaryngol. 2009 Feb;129(2):195-8. doi: 10.1080/00016480802078101. PMID 18607926
- [Background] Blomgren K, Qvarnberg YH, Valtonen HJ. A prospective study on pros and cons of electrodissection tonsillectomy. Laryngoscope. 2001 Mar;111(3):478-82. doi: 10.1097/00005537-200103000-00018. PMID 11224779
- [Background] Gysin C, Dulguerov P. Hemorrhage after tonsillectomy: does the surgical technique really matter? ORL J Otorhinolaryngol Relat Spec. 2013;75(3):123-32. doi: 10.1159/000342314. Epub 2013 Aug 22. PMID 23978795
- [Background] Juul MLB, Rasmussen ER, Howitz MF. Incidence of post-tonsillectomy haemorrhaging in Denmark. Dan Med J. 2020 Aug 1;67(8):A11190640. PMID 32741442
- [Background] Soderman AC, Odhagen E, Ericsson E, Hemlin C, Hultcrantz E, Sunnergren O, Stalfors J. Post-tonsillectomy haemorrhage rates are related to technique for dissection and for haemostasis. An analysis of 15734 patients in the National Tonsil Surgery Register in Sweden. Clin Otolaryngol. 2015 Jun;40(3):248-54. doi: 10.1111/coa.12361. PMID 25515059
- [Background] Lowe D, van der Meulen J; National Prospective Tonsillectomy Audit. Tonsillectomy technique as a risk factor for postoperative haemorrhage. Lancet. 2004 Aug 21-27;364(9435):697-702. doi: 10.1016/S0140-6736(04)16896-7. PMID 15325834
- [Background] Wulu JA, Chua M, Levi JR. Does suturing tonsil pillars post-tonsillectomy reduce postoperative hemorrhage?: A literature review. Int J Pediatr Otorhinolaryngol. 2019 Feb;117:204-209. doi: 10.1016/j.ijporl.2018.12.003. Epub 2018 Dec 4. PMID 30611028